CLINICAL TRIAL: NCT03778736
Title: Can Cumulase Reduce the Shear Stress During Denudation for ICSI Cycles of ≤ 8 Cumulus-oocytes Complexes
Brief Title: Using Cumulase for Denudation of Cycles With ≤ 8 Cumulus-oocytes Complexes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banoon IVF Center (Other); Quena IVF Center (Unknown)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IbnSina-Cumulase
Record Dates: First submitted 2018-12-15; First posted 2018-12-19 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cumulase denudation (Experimental)
  Interventions: Other: Cumulase denudation
- Hyaluronidase denudation (No Intervention)

INTERVENTIONS:
Other: Cumulase denudation — Testing the effect of cumulase for women with poor oocyte yield due to poor ovarian reserve
  Arms: Cumulase denudation

SUMMARY:
The cumulus-corona-oocyte complex (COCs) surrounds each oocyte and must be removed prior to intracytoplasmic sperm injection (ICSI). This is traditionally achieved with a bovine-derived hyaluronidase followed by mechanical denudation through pipetting. A human recombinant hyaluronidase (Cumulase) has been developed to circumvent the problems and concerns associated with the animal origin and lack of purity of the bovine-derived form of the enzyme. whether cumulase offers a higher chance for success after ICSI for women with 8 COCs or lower remains an open question.

ELIGIBILITY:
Inclusion Criteria:

* ICSI indicated partcipants

Exclusion Criteria:

* severe medical disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 586 (Actual)
Dates: Start 2018-01-27 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 16 weeks
  Continued pregnancy after 12 weeks of gestation

SECONDARY OUTCOMES:
Biochemical pregnancy | Two weeks
  Positive b-hCG at two weeks or more after embryo transfer
Clinical pregnancy rate | 7 weeks
  Detection of gestational sac with a heartbeat on ultrasound at 7 weeks of gestation
Embryo developmental rate | 6 days of culture
  fertilized oocytes per injected oocytes and developed embryos per fertilized oocytes

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Qena Fertility Center, Qina, Qena Governorate
  - Banon Assiut, Asyut
  - IbnSina IVF Center, Sohag

IPD SHARING:
Plan to Share IPD: No